CLINICAL TRIAL: NCT03124238
Title: Effect of Massage Therapy on Muscle Fatigue in Individuals With Low Back Pain: Physiological or Clinical Changes
Brief Title: Effect of Massage Therapy on Muscle Fatigue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université du Québec à Trois-Rivières (Other)
Responsible Party: Principal Investigator, Martin Descarreaux, Professor, Université du Québec à Trois-Rivières
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: UQTR-2016-MASSO
Record Dates: First submitted 2017-04-11; First posted 2017-04-21 (Actual); Last update posted 2017-04-24 (Actual); Status verified 2017-04

CONDITIONS: Low Back Pain
Keywords: massage
MeSH Terms: conditions — Low Back Pain | interventions — Massage

STUDY DESIGN:
Intervention Model Description: repeated measures crossover
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Massage (Experimental): Massage therapy of the lumbar muscles in a prone position during 30 minutes
  Interventions: Other: Massage
- Control (No Intervention): Rest during 5 minutes in a prone position

INTERVENTIONS:
Other: Massage — Massage therapy localized to the back of the individuals for a duration of 30 minutes
  Arms: Massage

SUMMARY:
The main objective of the current proposal is to investigate the clinical and physiological changes triggered by massage therapy in a group of individuals with chronic low back pain experiencing muscular fatigue.

The investigators believe these objectives are in line with the "2014 Massage Therapy Research Fund research priorities", since the results produced by these investigations will generate knowledge with regard to the short term clinical efficacy of massage therapy and will provide critical information related to the physiological mechanisms underlying massage therapy clinical effects. Most importantly, the combined assessment of clinical and physiological outcomes will also yield key information to identify specific biological components of the massage therapy intervention. Determining the presence of a biological mechanism is, as for any treatment, considered one of the necessary criteria to declare a causal relationship between a specific intervention and its associated clinical effects. The investigators strongly believe that the proposed research will contribute to the identification of specific mechanisms that will complement the emerging clinical evidence supporting massage therapy in the treatment of chronic low back pain.

The proposed research project will involve researchers and future practitioners of massage therapy. In conjunction with a high quality research environment, it is the goal of the investigators to create an educational environment for undergraduate and graduate students that will foster interdisciplinary collaboration in order to ensure a diversified; high quality training of young researchers and clinician scientists working in the field of manual therapies.

ELIGIBILITY:
Inclusion Criteria:

* Non specific low back pain

Exclusion Criteria:

* Low back pain of specific origin including but not limited to:

herniated disk fractures spondylolisthesis

* inflammatory rheumatic disease
* infectious disease
* neuromuscular disease
* vascular disease
* connective tissue disease
* severe disabling pain
* neurologic signs and symptoms
* pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2016-11-01 (Actual); Study Completion 2016-11-01 (Actual)

PRIMARY OUTCOMES:
Median frequency slope of the lumbar muscles (Hz/s) | assessed immediatly after massage or rest
  Fatigue will be assess during a extensor muscle endurance task throught surface electromyography electrodes (the more the slope value is negative and high, the more the muscle presents an important fatigue)
Maximal isometric force of the lumbar muscles (Newtons) | assessed immediatly after massage or rest
  Back extensor isometric force is assess throught surface electromyography electrodes during a five seconds maximal volontary contraction

CONTACTS AND LOCATIONS:
Overall Officials: Martin Descarreaux, DC PhD, Principal Investigator — Université du Québec à Trois-Rivières

IPD SHARING:
Plan to Share IPD: No
No data sharing will be done